CLINICAL TRIAL: NCT04764370
Title: Guo's Aortic Arch Reconstruction: The First in Man Study of WeFlow-Arch Modular Embedded Branch Stent Graft System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WeFlow-Arch V1.0
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Aortic Arch; Aneurysm, Dissecting
Keywords: Aortic Arch; Aneurysm; Dissecting; Ulcers
MeSH Terms: conditions — Aneurysm; Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WeFlow-Arch Moduler Embedded Branch Stent Graft System (Experimental)
  Interventions: Device: WeFlow-Ach Moduler Embedded Branch Stent Graft System

INTERVENTIONS:
Device: WeFlow-Ach Moduler Embedded Branch Stent Graft System — The modular embedded aortic arch stent graft system consists of the embedded ascending aorta stent graft system, the arch aorta stent graft system and the branch stent system.

SUMMARY:
This study is the first in man study of WeFlow-Arch Module Embedded Aorta Arch Stent Graft System

DETAILED DESCRIPTION:
The WeFlow-Arch Moduler Embedded Aorta Arch Stent Graft System first in man study is a prospective, single center, single arm trial, which will enroll a total of 20 patients. The goal of this study is to evaluate the safety and efficacy of WeFlow-Arch Moduler Embedded Aorta Arch Stent Graft System in the treatment of patients with lesions of the aortic arch.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 85 years old；
2. Diagnosed with aortic arch lesions requiring intervention, including true aortic arch aneurysms, pseudo-aortic arch aneurysms, dissection and ulcers involving the aortic arch;
3. The length of the ascending aorta is greater than 4cm (from the junction of the aortic sinus tube to the proximal edge of the innominate artery)；
4. Ascending aorta diameter ≥24mm and ≤44mm；
5. The diameter of the iliac artery ≥7mm ；
6. The diameter of the innominate artery ≤24mm, and the length ≥20mm；
7. Patients able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the subject him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol.

Exclusion Criteria:

1. Patients with ascending aortic aneurysm, dissection, ulcer, hematoma；
2. Experienced systemic infection during past three months;
3. History of aortic valve repair or replacement；
4. History of aortic surgery or endovascular repair surgery；
5. Carotid artery is severely narrowed, calcified, clotted, twisted；
6. Right axillary artery is severely narrowed, calcified, thrombosis, twisted；
7. Heart transplant；
8. Suffered MI or stroke during past three months；
9. Class IV heart function (NYHA classification)；
10. Pregnant or breastfeeding；
11. Allergies to contrast agents；
12. Life expectancy less than 12 months。

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Rate of no major adverse events related to device or surgery | 30 days after surgery
  Major adverse events related to device or surgery include: stroke, respiratory failure, pericardial tamponade, dissection or aneurysm rupture, paraplegia, stent occlusion, stent bend, stent displacement, thrombosis or rupture of the approach vessel, switch to open surgery, death, etc.

SECONDARY OUTCOMES:
Technical success rate | immediately after the surgery
  Successful delivery of the stent graft conveyors to their predetermined positions, accurate positioning and successful deployment of the stent, safe removal of the delivery device outside the body.
Immediate surgery success rate | immediately after the surgery
  Successful delivery of the stent graft, no major adverse events related to devices or surgery.
The clinical success rate | 12 months after the surgery
  Clinical success rate：12 months after the operation, there was no displacement of the stent, I and III endoleak requiring treatment, aneurysm enlargement or rupture, and branch stent occlusion.
The incidence rate of secondary operations within 12 months after surgery | 12 months after surgery
  The incidence rate of secondary operations within 12 months after surgery.
Adverse event rate within 12 months after surgery | 12 months after surgery
  Adverse event rate within 12 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No